CLINICAL TRIAL: NCT00574171
Title: A Phase II Trial of Lapatinib and Capectiabine for Patients With Refractory Advanced Colorectal Adenocarcinoma (LAP109859)
Brief Title: Phase II Trial of Lapatinib & Capecitabine for Patients With Refractory Advanced Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO 07201; A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); LAP109859 (Other Grant/Funding Number: Glaxo Smith Kline); NCI-2011-00477 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2016-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: lapatinib — 1250mg by mouth daily one hour before or after breakfast on a continuous basis.
  Other Names: Tykerb
Drug: Capecitabine — 2000mg/m2 of body surface area (BSA), by mouth, divided into twice daily dosing. Capecitabine will be given for days 1 through 14 of a 21 day cycle.
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to find out how effective this combination is as a second line treatment for colorectal cancer that has spread from one part of the body to another (metastasized) or has not metastasized but is considered inoperable (unable to be removed by surgery). The side effects and survival experienced by subjects receiving these drugs will also be evaluated. This is a phase II research study.

DETAILED DESCRIPTION:
1. To evaluate the response rate of lapatinib and capecitabine combination in patients with metastatic colon or rectal cancer.
2. To evaluate the toxicity and tolerability of lapatinib and capecitabine in this population.
3. To determine overall survival and disease free survival of lapatinib and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Pathologically confirmed, locally advanced or metastatic adenocarcinoma of the colon or rectum
* Patients must have had progression of disease on prior therapy with an oxaliplatin-containing or irinotecan containing regimen
* Proper radiographic documentation of measurable disease using RECIST criteria
* ECOG performance status (PS) of 0 or 1
* Laboratory parameters:

Hgb: ≥ 9.0 g/dl ANC ≥ 1500/ul Platelet ≥ 100,000/ul Creatinine ≤ 2x ULN OR Creatinine clearance ≥ 30 mg/ml Bilirubin ≤ 2x ULN AST ≤ 2x ULN or 5X ULN if liver metastases are present

* Patient has signed informed consent
* Toxicities from prior therapy (except alopecia and neuropathy) must have resolved to grade 1 or better prior to enrollment

Exclusion Criteria:

* Administration of more than one prior systemic chemotherapy for metastatic disease
* Pregnant or breast-feeding women: female patients must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. All at-risk female patients must have a negative serum pregnancy test within 7 days prior to randomization.
* Active inflammatory bowel disease, significant bowel obstruction, or chronic diarrhea (grade 2).
* Known human immunodeficiency virus (HIV) positivity or acquired-immunodeficiency-syndrome (AIDS)-related illness.
* No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer for which the patient has been disease-free for 3 years.
* Known CNS metastases
* Prior therapy which specifically and directly targets the EGFR pathway
* Significant history of uncontrolled cardiovascular disease, defined as:

  * History of uncontrolled or symptomatic angina
  * History of arrhythmias requiring medications, or clinically significant, with the exception of asymptomatic atrial fibrillation requiring anticoagulation
  * Myocardial infarction < 6 months prior to study entry
  * Cerebrovascular accident <6 months prior to study entry
  * Uncontrolled or symptomatic congestive heart failure
  * Ejection fraction below the institutional normal limit
  * Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcee J Jumonville, M.D., Study Chair — Gunderson Lutheran - LaCrosse
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lapatinib and Capecitabine: Capecitabine : 2000mg/m2 of body surface area (BSA), by mouth, divided into twice daily dosing. Capecitabine will be given for days 1 through 14 of a 21 day cycle.
  lapatinib : 1250mg by mouth daily one hour before or after breakfast on a continuous basis.
Period: Overall Study
Arm/Group | Lapatinib and Capecitabine
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Capecitabine : 2000mg/m2 of body surface area (BSA), by mouth, divided into twice daily dosing. Capecitabine will be given for days 1 through 14 of a 21 day cycle.
  lapatinib : 1250mg by mouth daily one hour before or after breakfast on a continuous basis.
Arm/Group | Arm 1
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Lapatinib/Capecitabine.
Time Frame: duration of study; on average 1 year
Measure: Number; unit: participants
Groups:
- Lapatinib/Capecitabine: lapatinib: 1250mg by mouth daily one hour before or after breakfast on a continuous basis. Capecitabine: 2000mg/m2 of body surface area (BSA), by mouth, divided into twice daily dosing. Capecitabine will be given for days 1 through 14 of a 21 day cycle.
Arm/Group | Lapatinib/Capecitabine
Number analyzed (Participants) | 29
participants
  PD | 4
  SD | 1

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=29)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (2)
Obstruction - small bowel, NOS (Gastrointestinal disorders) | 1 (2)
Death (General disorders) | 2 (2) — Death not associated with CTCAE term - Death NOS
Hypoxia (Cardiac disorders) | 1 (1) — related to patient's pulmonary embolism
Infection with normal ANC or Grade 1 or 2 neutrophils - Rectum - Presacral mass (Gastrointestinal disorders) | 1 (1)
Sedation from narcotic over dose. (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No